CLINICAL TRIAL: NCT05478018
Title: Type 1 Interferon Induced Changes to Exercise Adaptations in Systemic Lupus
Brief Title: Type 1 Interferon Induced Changes to Exercise Adaptations in Systemic Lupus Erythematosus Patients
Acronym: LUPEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Lupus and Vasculitis Clinic, Center for Rheumatology and Spine Diseases, Rigshospitalet (Unknown)
Responsible Party: Principal Investigator, Malte Lund Adamsen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-21039032
Record Dates: First submitted 2022-07-21; First posted 2022-07-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus; Interferon Deficiency
Keywords: Cardiac adaptations; Metabolic adaptations; High intensity interval training; Interleukin-6 signature; Tumor necrosis factor signature; Interferon signature
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — High-Intensity Interval Training; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The patients will be randomized to 12-week supervised exercise training intervention or no exercise training. The exercise training program includes three supervised sessions per week over a 12-week period.
  The program consists of high intensity endurance training on ergometer bicycles. The intensity will progress throughout the 12 weeks of training. The training consists of 10 minutes of warm up at 40-60% maximum heart rate (HRmax), followed by 25 minutes of high intensity interval training (4 bouts of 4 min at >85% HRmax interspaced by 3 minutes of low intensity training at 40-60% Hrmax) and finally a 3-10 min cool-down of 50% Hrmax
  Interventions: Behavioral: High Intensity Interval Training (HIIT)
- Non-Exercise (No Intervention): Control group, therefore no supervised exercise regime. Subjects are asked to not increase habitual exercise routines.

INTERVENTIONS:
Behavioral: High Intensity Interval Training (HIIT) — Supervised high-intensity interval training for 12 weeks three times per week
  Other Names: Aerobic Exercise
  Arms: Exercise

SUMMARY:
Investigating the physiological effects of the interferons type 1 and 2 (IFNs), and the cytokines Interleukin 6 (IL-6) and tumor necrosis factor (TNF) on the adaptive changes to exercise in patients with systemic lupus erythematosus (SLE).

The investigators hypothesize that the pathogenic blockage of IL-6 signalling that occurs in SLE, will decrease the cardiac and metabolic adaptations to aerobic exercise, and this decrease can be related to the IFN signature.

55 patients was included in a 12-week investigator blinded 1:1 randomised high intensity aerobic exercise intervention study.

DETAILED DESCRIPTION:
55 patients with SLE have been included and randomized in a 1:1 fashion to a 12 week high intensity interval training (HIIT) course or standard care.

Randomization was stratified by sex.

All patients will undergo baseline and followup testing including: VO2Max, Pulmonary Function, Capillaroscopy, OGTT, Blood Tests, Epigenetic Markers of IFN, TNF and IL-6 signalling, Echocardiography,DXA, Medical Examination, Acute Exercise Bout with blood tests during and after an exercise bout similar to the intervention. A subgroup of patients will be offered a 82-Rb Pet CT of the heart as opt-in.

The exercise programme consists of 12 weeks of tri-weekly exercise bouts of 38-45 minutes, following warm-up subjects will undergo 4 sets of 4 minute high intensity exercise, measured as the pulse being above 85% of HRmax for more than half the time; and 3 minute low to medium intensity exercise between the high intensity sets, measured as the pulse being between 40 to 60% of HRmax.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years by inclusion.
* Able to provide informed consent.
* Diagnosed SLE and fulfilling the classification criteria for SLE based on the American College of Rheumatology/EULAR criteria (SLICC)

Exclusion Criteria:

* Health conditions that prevent participating in the exercise intervention determined by the Research Coordinator these include but are not limited to

  * Major bone fracture at inclusion
  * Significant myalgias exacerbated by physical exercise
  * Active infectious disease such as Covid-19
  * Severe symptomatic pleuritis or pericarditis
* Corticosteroid use > 10mg/day at baseline
* Diagnosed with diabetes mellitus by physician
* Pregnancy
* SLEDAI-2k (with the SELENA modifications to Proteinuria changes so as to not exclude patients with chronic proteinuria) > 10
* Contraindications to 82Rb-PET with adenosine stress (according to local guidelines at the Dept. of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, which are in accordance with the recommendations of the European Association of Nuclear Medicine)

  * Fever, myocarditis or endocarditis
  * Previous heart transplantation
  * Dysregulated atrial or ventricular tachyarrhythmias
  * Severe chronic obstructive pulmonary disease with a FEV1 of less than 50% of predicted
  * Second or third degree sinoatrial or atrioventricular block
  * Active bronchospasm at the time of the scan
  * Systolic blood pressure <90 or >200 mmHg at the time of the scan
  * Treatment with theophyllin within 7 days of the scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in maximal aerobic capacity (VO2max) | 12 weeks
  Measured by VO2max test
Patient reported Fatigue | 12 weeks
  measured by Fatigue Severity Scale Questionnaire (FSS)

SECONDARY OUTCOMES:
Y2K updated SLE disease activity (SLEDAI-2K) with the SELENA modifications | 12 weeks
  Physician evaluated changes in measures of SLE on a scale of 0-105 encompassing symptoms from 9 organs, higher scores indicate increased disease activity.
Short Form (SF)-36 Health Survey (0-100) | 12 weeks
  Patient reported outcome measures (PROMs), Possible scores range from 0 to 100, with higher scores representing better health status
Change in Epigenetic Expression related to IFN alpha | 12 weeks
  Measured by mRNA analysis

OTHER OUTCOMES:
Systemic Lupus Erythematosus Disease Activity Index 2000 Responder Index-50 (SRI-50) | 12 weeks
  Itemized Physician evaluated changes in measures of SLEDAI-2K on a scale from 0-22 that account for partial improvements in condition, higher scores indicate increased disease activity.
Visual Analog Scale (VAS) of global disease by Physician (0-100%) | 12 weeks
  Physician evaluated changes in measures of SLE (0-100% of line segment), higher scores equal higher disease activity (worse)
Visual Analog Scale (VAS) fatigue (0-100) | 12 weeks
  Patient reported outcome measures (PROMs) , higher scores equal higher fatigue (worse)
Visual Analog Scale (VAS) pain (0-100) | 12 weeks
  Patient reported outcome measures (PROMs), higher scores equal more pain (worse)
SLAQ - (range 0 -33) | 12 weeks
  Patient reported outcome measures (PROMs), Possible scores range from 0 to 33, with higher scores representing more active SLE (worse)
SLE activity Visual Analog Scale - (1-10) | 12 weeks
  Patient reported outcome measures (PROMs), Possible scores range from 1 to 10, with higher scores representing more active SLE
Proteinuria | 12 weeks
  Measured by Dipstick in a semiquantitive manner with the following categories indicating increased concentration, negative, +/-, 1+, 2+, 3+, 4+.
Body composition - Total adipose tissue - Weight | 12 weeks
  Measured by DXA Scan - fat(g)
Body composition - Total adipose tissue - Percentage | 12 weeks
  Measured by DXA Scan - fat(%)
Body composition - Android adipose tissue - Weight | 12 weeks
  Measured by DXA Scan - android fat(g)
Body composition - Android adipose tissue - Percentage | 12 weeks
  Measured by DXA Scan - android fat(%)
Body composition - Gyneoid adipose tissue - Weight | 12 weeks
  Measured by DXA Scan - Gyneoid fat(g)
Body composition - Gyneoid adipose tissue - Percentage | 12 weeks
  Measured by DXA Scan - Gyneoid fat(%)
Body composition - Total Lean Mass - Weight | 12 weeks
  Measured by DXA Scan - Muscle Mass(g)
Body composition - Bone Mass Density - Weight/square-centimeter | 12 weeks
  Measured by DXA Scan - BMD(g/cm^2)
Waist-To-Height Ratio | 12 weeks
  measured with tape measure
Dynamic Spirometry - Forced Expiratory Volume at 1 second (FEV1) volume | 12 weeks
  Pulmonary function testing, FEV1 volume
Dynamic Spirometry - Forced Expiratory Volume at 1 second (FEV1) Percent of expected | 12 weeks
  Pulmonary function testing, FEV1%
Dynamic Spirometry - Forced Vital Capacity Volume | 12 weeks
  Pulmonary function testing, FVC Volume
Dynamic Spirometry - Forced Vital Capacity - Percent of Expected | 12 weeks
  Pulmonary function testing FVC%
Dynamic Spirometry Forced Expiratory Volume at 1 second (FEV1) by Forced Vital Capacity - Ratio | 12 weeks
  Pulmonary function testing, FEV1/FVC ratio
Dynamic Spirometry Forced Expiratory Volume at 1 second (FEV1) by Forced Vital Capacity - Ratio - Percentage of expected | 12 weeks
  Pulmonary function testing, FEV1/FVC ratio %
Dynamic Spirometry - Total Lung Capacity - Volume | 12 weeks
  Pulmonary function testing, TLC Volume
Dynamic Spirometry - Total Lung Capacity - Percentage of expected | 12 weeks
  Pulmonary function testing, TLC%
Dynamic Spirometry - Residual Volume - Volume | 12 weeks
  Pulmonary function testing, RV-Volume
Dynamic Spirometry - Residual Volume - Percentage of Expected | 12 weeks
  Pulmonary function testing, RV%
Dynamic Spirometry - Alveolar Volume - Volume | 12 weeks
  Pulmonary function testing, AV-Volume
Dynamic Spirometry - Alveolar Volume - Percentage of expected | 12 weeks
  Pulmonary function testing, AV-%
Dynamic Spirometry - Diffusing capacity for Carbon Monoxide - Volume | 12 weeks
  Pulmonary function testing, DLCOc-Volume
Dynamic Spirometry - Diffusing capacity for Carbon Monoxide - Percentage | 12 weeks
  Pulmonary function testing, DLCOc-%
Dynamic Spirometry - Carbon monoxide transfer coefficient - diffusing capacity per liter of lung volume | 12 weeks
  Pulmonary function testing, KCO-Volume
Dynamic Spirometry - Carbon monoxide transfer coefficient - diffusing capacity per liter of lung volume - percentage of expected | 12 weeks
  Pulmonary function testing, KCO-%
Oral glucose tolerance test | 12 weeks
  75g of glucose taken while fasting
Peripheral Capillary Changes - Capillary Density | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician (score of 1-4, higher scores equal fewer capillaries)
Peripheral Capillary Changes - Average Capillary Width (micrometers) | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician - Width Measured in µm
Peripheral Capillary Changes - Average Capillary Length(micrometers) | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician - Length Measured in µm
Peripheral Capillary Changes - Count of avascular areas | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician - Avascular Areas (1-4 higher scores indicate more avascular areas)
Peripheral Capillary Changes - Capillary Disorganization | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician - Capillary Disorganization (1-4 higher scores indicate more avascular areas)
Peripheral Capillary Changes - Microhemorrhages (average per finger) | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician - Microhemorrhages (avg per finger)
Peripheral Capillary Changes - Bushy Capillaries (average per millimeter) | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician - Bushy Capillaries (average per millimeter)
Peripheral Capillary Changes - Megacapillaries (average per millimeter) | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician - Megacapillaries (average per millimeter)
Peripheral Capillary Changes - Meandering capillaries (average per millimeter) | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician - Meandering capillaries (average per millimeter)
Peripheral Capillary Changes - Tortous capillaries (average per millimeter) | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician - Tortous capillaries (average per millimeter)
Peripheral Capillary Changes - Other Findings | 12 weeks
  Measured by Nailfold Capillaroscopy by trained physician - Physicians comment
Change in fasting total cholesterol, low-density lipoprotein (LDL)-cholesterol and high-density lipoprotein (HDL)-cholesterol (mmol/L). Following an overnight fast (10 hours) | 12 weeks
  blood samples are collected and processed by a trained laboratory technician and analysed according to standard procedures.monitors (AX3; Axivity, Newcastle upon Tyne, UK) for a 3 to 5 day period
Change in triglycerides (mmol/L). Following an overnight fast (10 hours) | 12 weeks
  blood samples are collected and processed by a trained laboratory technician and analysed according to standard procedures.monitors (AX3; Axivity, Newcastle upon Tyne, UK) for a 3 to 5 day period
left ventricular and atrial end-diastolic volume | 12 weeks
  measured by echocardiography
global longitudinal strain | 12 weeks
  measured by echocardiography
stroke volume | 12 weeks
  measured by echocardiography
left ventricular ejection fraction | 12 weeks
  measured by echocardiography
Left ventricular mass | 12 weeks
  measured by echocardiography
coronary perfusion reserve | 12 weeks
  measured by echocardiography (& 82Rb-PET-CT)
Myocardial blood flow | 12 weeks
  Measured by 82Rb-Pet-CT, on a subset of 40 participants
Axial accelerometer-based physical activity monitors | 12 weeks
  Free-living physical activity is measured using axial accelerometer-based physical activity monitors (AX3; Axivity, Newcastle upon Tyne, UK) for a 3 to 5 day period
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for High Sensitvity C-Reactive Protein | 12 weeks
  Analyzed for HS-CRP
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for Il-6 | 12 weeks
  Analyzed for Il-6
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for sIL-6r | 12 weeks
  Analyzed for soluble Il-6-receptor
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for Il-1 | 12 weeks
  Analyzed for Il-1
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for Il-10 | 12 weeks
  Analyzed for Il-10
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for IFNα | 12 weeks
  Analyzed for IFNα
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for IFNγ | 12 weeks
  Analyzed for IFNγ
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for hgb | 12 weeks
  Analyzed for hemoglobin
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for plates | 12 weeks
  Analyzed for thrombocytes
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for Na | 12 weeks
  Analyzed for sodium
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for K | 12 weeks
  Analyzed for potassium
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for Cl | 12 weeks
  Analyzed for chloride
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for hct | 12 weeks
  Analyzed for hematocrit.
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for Ferritin | 12 weeks
  Analyzed for ferritin
Change in peripheral blood Adaptation to Acute Exercise Bout - Analyzed for leucocyte differential | 12 weeks
  Analyzed for Leukocyte Differential
Change in Epigenetic Expression related to IFN Beta | 12 weeks
  Measured by mRNA analysis on PBMCs
Change in Epigenetic Expression related to IFN Gamma | 12 weeks
  Measured by mRNA analysis
Change in Epigenetic Expression related to TNF | 12 weeks
  Measured by mRNA analysis
Change in Epigenetic Expression related to IL-6 | 12 weeks
  Measured by mRNA analysis on PBMCs
Dietary Changes - Energy intake (kJ/day) | 12 weeks
  Patient Reported by dietary diary
Dietary Changes - carbohydrate intake (g/day) | 12 weeks
  Patient Reported by dietary diary
Dietary Changes - lipid intake (g/day) | 12 weeks
  Patient Reported by dietary diary
Dietary Changes - Protein intake (g/day) | 12 weeks
  Patient Reported by dietary diary
Dietary Changes - Other intake (categorical) | 12 weeks
  Patient Reported by dietary diary
Muscle Biopsy for epigenetic markers of inflammation and myokine signalling | 12 weeks
  Optional for Participants: mRNA expression of genes related to TNF, IL-6, IFN alpha, beta and Gamma signalling
Muscle Biopsy for epigenetic markers of physical activity | 12 weeks
  Optional for Participants: NF-κB p65 DNA binding activity (ELISA), phosphorylated and total JNK, phosphorylated AMPK (p-AMPK) total AMPK (Western blotting).
Muscle Biopsy for epigenetic markers of physical activity - NF-κB p65 DNA binding activity (ELISA) | 12 weeks
  Optional for Participants: NF-κB p65 DNA binding activity (ELISA) & NF-κB binding activity (Western blotting).
Muscle Biopsy for epigenetic markers of physical activity - c-Jun N-terminal kinase | 12 weeks
  Optional for Participants: phosphorylated and total JNK,
Muscle Biopsy for epigenetic markers of physical activity - AMP-activated protein kinase | 12 weeks
  Optional for Participants: phosphorylated AMPK (p-AMPK) total AMPK (Western blotting).
Autonomic Nerve Function Test - Resting HR by Vagus(tm) | 12 weeks
  Resting heart rate measured by R-R intervals on 1-lead ECG
Autonomic Nerve Function Test - Rise from supine ratio of RR by Vagus(tm) | 12 weeks
  Rise from supine ratio of R-R intervals on 1-lead ECG
Autonomic Nerve Function Test - Expiration Inspiration ratio of RR by Vagus(tm) | 12 weeks
  Expiration/Inspiration ratio of R-R intervals on 1-lead ECG
Autonomic Nerve Function Test - Valsalva Maneuver ratio of RR by Vagus(tm) | 12 weeks
  Valsalva Maneuver ratio of R-R intervals on 1-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Ronan Martin G Berg, MD, DMSc, Study Chair — Center for Physical Activity Research; Iben E Rasmussen, MSc, Study Chair — Center for Physical Activity Research; Simon Jønck, MD, Study Chair — Center for Physical Activity Research; Malte L Adamsen, MD, Principal Investigator — Center for Physical Activity Research
Locations (1):
- Center for Physical Activity Research, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study will be made publicly available 6 months after first publication. Academic researchers with interest in systemic lupus erythematosus or exercise therapy can contact the authors to get access before this embargo.
  Data or samples shared will be coded, with no PHI included.
  Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted immediate upon publication of the first paper, 6 months after article publication anonymized data will be made publicly accessible.
  All data shared will be done in a fully anonymized way.
Access Criteria: Access for the first 6 months following publication can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
  Following the first 6 months anonymized data will be publicly available.
  For more information or to submit a request, please contact Malte.Lund.Adamsen.02@regionh.dk or Soeren.Jacobsen.01@regionh.dk
URL: https://github.com/Malte-Lund

DOCUMENTS (2):
  • Study Protocol (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT05478018/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT05478018/SAP_001.pdf